CLINICAL TRIAL: NCT02688855
Title: Prospective, Randomized, Double-Blinded, Controlled Multi-Center Clinical Trial Evaluating the Use of Non-Invasive CMF Bone Stimulation as Adjunct to Surgical Treatment of Ankle Fractures
Brief Title: CMF Bone Stimulation as Adjunct to Surgical Treatment of Ankle Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Encore Medical, L.P. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PS-607
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Last update posted 2022-03-21 (Actual); Status verified 2021-12

CONDITIONS: Bimalleolar Ankle Fractures
Keywords: Bone Growth Stimulator; Ankle Fracture
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Investigational Group (Experimental): Standard Rigid Fixation + Active OL1000 device
  Interventions: Device: Active Combined Magnetic Field OL1000 Bone Growth Stimulator
- Control Group (Sham Comparator): Standard Rigid Fixation + Sham OL1000 device
  Interventions: Device: Sham Combined Magnetic Field OL1000 Bone Growth Stimulator

INTERVENTIONS:
Device: Active Combined Magnetic Field OL1000 Bone Growth Stimulator — Active CMF OL1000 Device
  Other Names: CMF OL1000
  Arms: Investigational Group
Device: Sham Combined Magnetic Field OL1000 Bone Growth Stimulator — Sham CMF OL1000
  Other Names: CMF OL1000
  Arms: Control Group

SUMMARY:
The OL1000 is intended to be used as a non-invasive adjunctive treatment for adult males or females that have sustained a closed, unstable ankle fracture that requires surgical treatment for stabilization. The initiation of the adjunctive treatment is to begin within 11 days of surgical stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Subject is diagnosed with an unstable, closed, isolated fracture of the ankle and underwent operative stabilization with plate(s) and/or screws (Weber Ankle Fracture Classification B and C)

Exclusion Criteria:

* Subject has an open fracture
* Subject has any additional fractures of another bone besides the ankle fracture that is to be treated in the study including the contralateral ankle
* Surgical stabilization was definitively performed with an external fixation system
* Surgical stabilization was performed in such a manner that it will result in a fusion of the ankle joint
* Malreduced Ankle as described by Phillips, et al 1985 JBJS
* Surgical procedure included the use of osteoinductive materials in addition to rigid fixation
* BMI ≥ 40 kg/m2

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2017-01-23 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change overtime of Olerud and Molander Ankle Score (OMAS) | 6 weeks, 8 weeks, 10 weeks and 12 weeks
Non-powered, composite safety endpoint consisting of: Joint Position Outcome Radiographic Failure and Repeat, Unplanned Surgery at the Operative Site and Device-Related Serious Adverse Events | 6 months & 12 months

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - University of Arizona, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Orthopaedic Associates of South Broward, P.A., Hollywood, Florida
  - OrlandoHealth, Orlando, Florida
  - William Beaumont Hospital, Royal Oak, Michigan
  - Rutgers Biomedical Health Sciences, Newark, New Jersey
  - University of Rochester, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Phillips WA, Schwartz HS, Keller CS, Woodward HR, Rudd WS, Spiegel PG, Laros GS. A prospective, randomized study of the management of severe ankle fractures. J Bone Joint Surg Am. 1985 Jan;67(1):67-78. PMID 3881447
- [Result] Olerud C, Molander H. A scoring scale for symptom evaluation after ankle fracture. Arch Orthop Trauma Surg (1978). 1984;103(3):190-4. doi: 10.1007/BF00435553. PMID 6437370
- See also: Related Info — http://www.djoglobal.com/products/cmf/cmf-ol1000